CLINICAL TRIAL: NCT03587428
Title: In-house Study to Determine the Effect of Two Zinc-containing Toothpaste Formulations on Viability of Bacteria in Saliva
Brief Title: Effect of Two Toothpastes on Bacteria in Saliva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202287
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-04

CONDITIONS: Oral Health
MeSH Terms: interventions — Mineral Waters

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zinc-A toothpaste (Experimental): In this arm, participants received Zinc-A toothpaste (test product 1) in the form of slurry.
  Interventions: Drug: Zinc-A toothpaste
- Zinc-B toothpaste (Experimental): In this arm, participants received Zinc-B toothpaste (test product 2) in the form of slurry.
  Interventions: Drug: Zinc-B toothpaste
- Mineral Water (Other): In this arm, participants received mineral water.
  Interventions: Other: Mineral water

INTERVENTIONS:
Drug: Zinc-A toothpaste — Participants received 6.0 grams (g) [± 0.3g] of the Zinc-A toothpaste in the form of slurry, one day per treatment (with at least 2 [generally 7] days between treatments. Participants emptied the contents of the dosing cup into their mouth, swilled the product around their mouth for 2 timed minutes then they expectorated into a sink.
  Arms: Zinc-A toothpaste
Drug: Zinc-B toothpaste — Participants received 6.0 grams (g) [± 0.3g] of the Zinc-B toothpaste in the form of slurry, one day per treatment (with at least 2 [generally 7] days between treatments. Participants emptied the contents of the dosing cup into their mouth, swilled the product around their mouth for 2 timed minutes then they expectorated into a sink.
  Arms: Zinc-B toothpaste
Other: Mineral water — Participants received 6.0g (±0.3g) of mineral water (by weighing out), one day per treatment (with at least 2 [generally 7] days between treatments). Participants emptied the contents of the dosing cup into their mouth, swilled the product around their mouth for 2 timed minutes then they expectorated into a sink.
  Arms: Mineral Water

SUMMARY:
This study investigated the ability of two zinc-containing toothpaste formulations (Zinc A and Zinc B) to reduce the level of bacteria in saliva in the two-hour period after their use, compared to the effect of rinsing with water alone.

DETAILED DESCRIPTION:
This was a single centre, three treatment, randomized, blinded, cross-over study which involved rinsing with slurries of two sodium fluoride-silica dentifrices containing zinc chloride and sodium citrate, and with water alone. The study consisted of four Visits: Visit 1 (Screening), Visit 2 (Treatment 1), Visit 3 (Treatment 2), Visit 4 (Treatment 3). There was a minimum two days wash out period before the first treatment visit and between treatment visits to avoid any treatment carry-over effect. During that time participants brushed as normal (twice-daily) at home with a washout toothpaste and a toothbrush which was provided at screening. Participants were required not to brush their teeth on the morning of the treatment visits and not to eat or drink for 2 hours prior to the treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Personnel: GSKCH permanent and contract/contingency workers.
* Consent: Demonstrated understanding of the study and was willing to participate and had received a signed and dated copy of the informed consent form.
* Compliance: Understood, was willing and able and complied with all study procedures and restrictions.
* General Health: Good general health
* Oral Health: Good oral health
* Salivary Flow Rate: Had a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2milliliter per minute (ml/min); stimulated whole saliva flow rate ≥ 0.8ml/min)

Exclusion Criteria:

* Study personnel: Members of the clinical study staff.
* Pregnancy: Pregnant Women
* Breast-feeding: Women who were breast-feeding.
* Allergy/Intolerance: Had Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Medication: a) Used an antimicrobial mouthwash within 48 hours of the test visit e.g. Listerine, Corsodyl etc. b) had taken, antibiotics within 2 weeks of the test visit.
* Oral Surgery and Dental Conditions: a)Had an on-going dental treatment b) Had any oral surgery or extraction within 6 weeks of screening c) Symptoms of oral pain or any self-reported oral ulcers or herpetic lesions
* Clinical Study Participation: a) Participation in a clinical study where they received an investigational drug within 2 weeks of the screening visit b) Previously participated in this study.
* Substance Abstinence: Participant who were unwilling to abstain from smoking for at least 2 hours prior to treatment visits.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2014-11-27 (Actual); Study Completion 2014-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Weybridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were recruited from one center in United Kingdom.
Pre-assignment Details: A total of 16 participants were screened, out of which 1 did not met the study criteria. Total of 15 participants were randomized to study treatments.
Groups:
- B-C-A: In this arm, participants received toothpaste in the form of slurry. The flow of events were first product B, then product C followed by product A, where, A is Zinc-A toothpaste, B is Zinc-B toothpaste and C is water.
- C-B-A: In this arm, participants received toothpaste in the form of slurry. The flow of events were first product C, then product B followed by product A, where, A is Zinc-A toothpaste, B is Zinc-B toothpaste and C is water.
- A-B-C: In this arm, participants received toothpaste in the form of slurry. The flow of events were first product A, then product B followed by product C, where, A is Zinc-A toothpaste, B is Zinc-B toothpaste and C is water.
- C-A-B: In this arm, participants received toothpaste in the form of slurry. The flow of events were first product C, then product A followed by product B, where, A is Zinc-A toothpaste, B is Zinc-B toothpaste and C is water.
- B-A-C: In this arm, participants received toothpaste in the form of slurry. The flow of events were first product B, then product A followed by product C, where, A is Zinc-A toothpaste, B is Zinc-B toothpaste and C is water.
- A-C-B: In this arm, participants received toothpaste in the form of slurry. The flow of events were first product A, then product C followed by product B, where, A is Zinc-A toothpaste, B is Zinc-B toothpaste and C is water.
Period: Period 1
Arm/Group | B-C-A | C-B-A | A-B-C | C-A-B | B-A-C | A-C-B
Started | 3 | 2 | 3 | 3 | 2 | 2
Completed | 3 | 2 | 3 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | B-C-A | C-B-A | A-B-C | C-A-B | B-A-C | A-C-B
Started | 3 | 2 | 3 | 3 | 2 | 2
Completed | 3 | 2 | 3 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | B-C-A | C-B-A | A-B-C | C-A-B | B-A-C | A-C-B
Started | 3 | 2 | 3 | 3 | 2 | 2
Completed | 3 | 2 | 3 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants completed the study and were included in the safety and intent-to-treat (ITT) populations. All efficacy analyses were conducted on the ITT population.
Groups:
- Overall: Includes participants that were given interventions: Zinc-A toothpaste or Zinc-B toothpaste or Mineral Water
Arm/Group | Overall
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Area Under the Curve Between 0 and 2 Hours (AUC [0-2] Hours) for Total Viable Counts (TVCs) of Bacteria in Saliva Using Traditional Plating Technique
Description: Area Under the Curve (AUC) between 0 and 2 hours (hr) was assessed using traditional plating technique which provides the total viable counts (TVCs) of anaerobic bacteria. This outcome measure is AUC of change from baseline in log TVC. AUC for each time-point were calculated individually for each participant for each treatment and were aggregated into an AUC measurement. The aggregated AUC measurement was calculated in the order that first the collected data is logged which is further analyzed by change in log. Then, AUC 0-2hr change in log was calculated using the trapezoidal rule. The resulted values were then divided by 2hr to take out time units and are logged to calculate bacteria count. Hence, the outcome measure calculates change from baseline in log10-transformed AUC 0-2hr over the range from pre-treatment time point (0hr) to the concentration at 120 minutes (min) i.e., 2hr.
Time Frame: Change from baseline in log10-transformed AUC 0-2hr
Population: The efficacy analysis was performed on Intent to Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Log10 (cells/ml)
Arm/Group | Zinc-A Toothpaste | Zinc-B Toothpaste | Mineral Water
Number analyzed (Participants) | 15 | 15 | 15
Log10 (cells/ml)
  At Baseline | 8.818 (1.3909) | 8.785 (1.3643) | 8.845 (0.7271)
  Change from Baseline in AUC at 120 minutes | -0.037 (2.4945) | -0.348 (2.8109) | 0.193 (1.6106)
Statistical Analysis 1: Comparison: Zinc-A Toothpaste vs Mineral Water; Test type: Superiority; p = 0.1787, ANCOVA; ANCOVA for treatment and period as fixed effects and subject as random effect and two baseline terms as covariates; Mean Difference (Final Values) = -0.3252, 95% CI 2-sided [-0.8101 to 0.1596] — Difference is first named treatment minus second named treatment; a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: Zinc-B Toothpaste vs Mineral Water; Test type: Superiority; p = 0.0063, ANCOVA; ANCOVA for treatment and period as fixed effects and subject as random effect and two baseline terms as covariates; Mean Difference (Final Values) = -0.7037, 95% CI 2-sided [-1.1886 to -0.2187] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in AUC (0-2) Hours for the Ratio of Live:Dead Bacteria Using Live-dead Staining Technique
Description: Anaerobic bacteria were counted using live:dead staining technique. Change from baseline in AUC (0-2)hr was calculated for the ratio of live and dead bacteria. Viable bacterial counts for each time-point were calculated individually for each participant for each treatment and were aggregated into an AUC measurement. AUC was calculated using the trapezoidal rule and using nominal time points. The resulted values were then divided by 2hr to take out time units. The AUC was calculated over the range from pre-treatment time point (0hr) to 2hr. In this outcome measure, the change from baseline is calculated in log ratio of live: dead.
Time Frame: Baseline up to 2 hours
Population: The efficacy analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: Ratio (unitless)
Arm/Group | Zinc-A Toothpaste | Zinc-B Toothpaste | Mineral Water
Number analyzed (Participants) | 15 | 15 | 15
Ratio (unitless)
  At Baseline | 0.758 (0.3961) | 0.946 (0.1495) | 0.906 (0.1856)
  Change from Baseline in AUC at 120 minutes | -7.612 (5.5419) | -10.927 (4.6267) | -1.024 (3.7681)

3. Secondary Outcome: Change From Baseline in log10-transformed Total Viable Bacterial Count Using Traditional Bacterial Plating Technique
Description: Anaerobic bacteria were counted using traditional plating technique. Total viable bacterial counts for each time-point was calculated individually for each participant for each treatment. Change from baseline in log 10 transformed total viable bacterial values was calculated.
Time Frame: At Baseline, 5 minutes, 15 minutes, 30 minutes, 1 hour and 2 hours post-treatment
Population: The efficacy analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: Log10 (cells/ml)
Arm/Group | Zinc-A Toothpaste | Zinc-B Toothpaste | Mineral Water
Number analyzed (Participants) | 15 | 15 | 15
Log10 (cells/ml)
  At 5 minutes | -0.364 (1.3410) | -0.474 (1.4832) | 0.144 (0.5679)
  At 15 minutes | -0.030 (1.2444) | -0.214 (1.5142) | 0.161 (0.9736)
  At 30 minutes | 0.092 (1.4285) | -0.130 (1.5997) | -0.177 (1.0780)
  At 1 hour | -0.032 (1.2486) | -0.175 (1.4857) | 0.193 (0.7781)
  At 2 hour | 0.009 (1.4097) | -0.129 (1.5035) | 0.127 (0.8379)

4. Secondary Outcome: Change From Baseline in Live:Dead Bacteria Ratio in Saliva Using Staining Technique
Description: Anaerobic bacteria were counted using live:dead staining technique. Change from baseline was calculated for the ratio of live to dead bacteria.
Time Frame: At Baseline, 30 minutes, 1 hour and 2 hours post-treatment
Population: The efficacy analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: Ratio (unitless)
Arm/Group | Zinc-A Toothpaste | Zinc-B Toothpaste | Mineral Water
Number analyzed (Participants) | 15 | 15 | 15
Ratio (unitless)
  At 30 minutes | -4.701 (3.3349) | -6.728 (2.7295) | -0.049 (1.8977)
  At 1 hour | -4.259 (3.1983) | -6.153 (2.6444) | -0.820 (2.4004)
  At 2 hour | -3.236 (3.1452) | -5.419 (2.6849) | -0.769 (2.7484)

ADVERSE EVENTS:
Time Frame: approximately 28 days
Description: All subjects who received treatment were included in the safety population. Adverse Events (AEs) were summarized by treatment group.
Arm/Group | Zinc-A Toothpaste | Zinc-B Toothpaste | Mineral Water
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.